CLINICAL TRIAL: NCT07068360
Title: Development and Validation of a Multimodal Physiotherapy Framework to Prevent and Mitigate Postural Hyperkyphosis in Postmenopausal Women: A Randomized Controlled Trial
Brief Title: Development and Validation of MPF to Prevent and Mitigate Postural Hyperkyphosis in Postmenopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PhDRSW/Batch-Fall23/2224
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hyperkyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Training +Postural Correction Exercises + Balance Training +Flexibility Exercises (Experimental)
  Interventions: Combination Product: Strength Training +Postural Correction Exercises + Balance Training +Flexibility Exercises
- Standard Intervention (Control Group) (Active Comparator)
  Interventions: Diagnostic Test: Standard Intervention (Control Group)

INTERVENTIONS:
Combination Product: Strength Training +Postural Correction Exercises + Balance Training +Flexibility Exercises — Interventions details (Group A) Strength Training Postural Correction Exercises Balance Training Exercises
  Flexibility Exercises:
  Arms: Strength Training +Postural Correction Exercises + Balance Training +Flexibility Exercises
Diagnostic Test: Standard Intervention (Control Group) — The control group will receive standard physiotherapy for postural hyperkyphosis.
  The standard intervention will consist of:
  Postural education: Educating participants on proper posture, body mechanics, and ergonomics in daily activities.
  Basic stretching exercises targeting the thoracic spine and back muscles. Recommendations for low-impact aerobics activities (e.g., walking or cycling) to promote overall healthThe standard intervention will be delivered over the same 12-week period, with two sessions per week. This group will not receive the integrated multimodal framework with strength training, postural correction, balance training, and flexibility exercises that the experimental group receives. Duration and Frequency
  Arms: Standard Intervention (Control Group)

SUMMARY:
Postural hyperkyphosis is common in postmenopausal women and leads to spinal dysfunction, pain, impaired balance, and increased fall risk. This study aims to develop and validate a multimodal physiotherapy framework to prevent and manage hyperkyphosis in this population. A randomized controlled trial will be conducted at Allied Hospital with 72 postmenopausal women aged 40-75 years, divided into intervention (multimodal physiotherapy with conventional care) and control (conventional care only) groups.

DETAILED DESCRIPTION:
The intervention includes strength, flexibility, postural correction, and balance training. The primary outcome is the change in Cobb's angle measured via radiographs; secondary outcomes include functional mobility and balance assessments using the Timed Up and Go Test, Berg Balance Scale, and Functional Reach Test. Data will be analyzed using SPSS v26. The study is expected to show significant improvements in spinal alignment, strength, balance, and reduced fall risk. The framework may offer a cost-effective, evidence-based approach for clinical and community rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 50-70 years.
* Kyphotic angle ≥40°, as measured by a flexicurve ruler or radiographic assessment.
* Postmenopausal for at least one year.
* Able to engage in rehabilitation exercises and follow instructions for physical activity..
* Living independently and capable of attending regular physiotherapy sessions.

Exclusion Criteria:

* Uncontrolled comorbidities such as cardiovascular disease, neurological disorders stroke or Parkinson's), or severe musculoskeletal conditions (e.g., advanced arthritis )
* History of spinal surgery within the last 6 months or spinal surgical implants. Severe osteoporosis (T-score < -2.5) and a history of multiple fractures.
* Pregnant or breastfeeding women. Cognitive impairments or mental health disorders that hinder adherence to the intervention.
* Inability to perform the exercises due to pain or disability.
* Participation in other rehabilitation or physiotherapy interventions for postural hyperkhyposis

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cobb's Angle | 18 Months
  Cobb's Angle is a radiographic measurement used to assess spinal curvature in conditions like hyperkyphosis and scoliosis. It is calculated by identifying the most tilted vertebrae at the top and bottom of the curve on an X-ray. Straight lines are drawn along their endplates, and perpendiculars from these lines intersect to form the Cobb's Angle. A normal thoracic kyphosis ranges from 20° to 40°, while angles exceeding 40° in adults or 50° in postmenopausal women indicate hyperkyphosis. Severe cases (>60°) may require medical intervention. Regular follow-ups help monitor treatment effectiveness in reducing spinal curvature.
Timed Up and Go (TUG) Test | 18 Months
  The TUG test assesses mobility, balance, and fall risk in older adults. The patient starts seated in a chair, stands up, walks 3 meters (10 feet), turns around, walks back, and sits down. The time taken to complete the task is recorded in seconds. A score of <10 seconds indicates normal mobility, 10-20 seconds suggests mild mobility impairment, and >30 seconds signifies a high fall risk and functional dependence. It is a simple, reliable tool commonly used in rehabilitation settings.
Berg Balance Scale (BBS) | 18 Months
  The BBS is a 14-item test used to assess balance and fall risk in older adults and neurological patients. Each task, such as standing on one foot or reaching forward, is scored from 0 to 4, with a total score of 56. A score of 41-56 indicates low fall risk, 21-40 suggests moderate risk, and ≤20 signifies a high risk of falls. The test is widely used due to its strong reliability and validity in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Faisalabad Medical University (Allied Hospital Faisalabad), Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No